CLINICAL TRIAL: NCT07222774
Title: Intention Interventions
Brief Title: Strengthening Intentions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 06281970
Record Dates: First submitted 2025-09-04; First posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-09

CONDITIONS: Influenza Vaccination; Behavior And Behavior Mechanism
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: We will compare the study outcomes between a control arm and the intervention arm.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): no intervention control arm, usual care
- intervention (Experimental): create, strengthen intention
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Experimental — behavioral intention
  Arms: intervention

SUMMARY:
participants are randomized to a study arm that measures intention to perform a health related behavior and follows up to measure behavior

ELIGIBILITY:
Inclusion Criteria: user of THEA -

Exclusion Criteria: non users of THEA

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
past behavior | 90 days
  whether behavior was performed

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States